CLINICAL TRIAL: NCT01850719
Title: Cost-effectiveness of Early Surgery Versus Conservative Treatment With Optional Delayed Meniscectomy in Older Patients. A Randomized Controlled Trial.
Brief Title: Early Surgery Versus Conservative Therapy for Meniscal Injuries in Older Patients
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Achmea Gezondheidszor (Other)
Responsible Party: Principal Investigator, Victor van de Graaf, MD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL4418.100.13
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Meniscal Tear
Keywords: Tibial meniscus; Arthroscopy; Meniscectomy; Conservative treatment; Physical therapy; Osteoarthritis knee joint
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic Partial Meniscectomy (Experimental)
  Interventions: Procedure: Arthroscopic Partial Meniscectomy
- Physical Therapy (Active Comparator)
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Procedure: Arthroscopic Partial Meniscectomy — Arthroscopic partial APM is performed within 4 weeks in day-care. No standard physical therapy is prescribed after surgery, as advised by the Dutch Orthopaedic Association Guidelines.
  Other Names: APM
  Arms: Arthroscopic Partial Meniscectomy
Other: Physical Therapy — Conservative treatment consist of 16 sessions PT and a home exercise program. These programs are developed for our population, 45-70 years, with a focus on closed-chain strength exercises and cardiovascular exercises.
  In case conservative treatment has failed, patients can cross-over and delayed APM is then performed. This can be done, from completion of the PT program, during the entire study.
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to determine the effectiveness of both arthroscopic knee surgery and physical therapy in the treatment of non-obstructive meniscal injuries in older patients.

The investigators assume equal improvement of physical function in both groups and reduced costs with conservative treatment.

DETAILED DESCRIPTION:
Rationale: Arthroscopic Partial Meniscectomy (APM) is the most performed orthopaedic procedure and is current standard treatment for patients with meniscal tears. Since superiority of APM over conservative treatment has not well been described and studies with direct comparison between APM and conservative treatment are sparse, therefore there is risk of large healthcare inefficiency.

Study design: Non-inferiority multicenter randomized controlled trial with an economic evaluation alongside. The study will be conducted by the Orthopaedic Research Consortium Mid-West Netherlands and performed in 6 clinics, including 2 academic medical centers.

402 patients between 45 and 70 years with Magnetic Resonance Imaging (MRI)-confirmed symptomatic, non-obstructive meniscal tears will be included. Patients will be assigned to either APM (n=201) or Physical Therapy (PT; n=201), with optional delayed APM (cross-over) when conservative treatment has failed. Block randomization will be done stratified for age and site. Data will be analysed on both intention to treat and per protocol basis.

Measurement points:

* Patients will be asked to complete questionnaires at baseline and 3, 6, 9, 12, 18, 24 and 60 months.
* At both 3 and 24 months they will visit the outpatient department for physical examination.
* At 24 and 60 months an X-ray will be obtained.

Sample size calculation: 402 patients, based on a power of 90%, an alpha of 0.05, a standard deviation of 20 points and a non-inferiority threshold of 8 points on the IKDC 'Subjective Knee Form'. Loss to follow up and cross-over have been taken into account in this calculation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 45 and 70 years of age at presentation.
* A meniscal tear visualized on MRI. The meniscal tear can either be isolated or combined with a partial asymptomatic Anterior Cruciate Ligament (ACL) injury or an asymptomatic degenerative ACL shown on MRI with no abnormal clinical findings (a negative Lachman test and Pivot Shift).
* Mental Competence.
* Willingness to comply with follow up schedule.
* Written informed consent.

Exclusion Criteria:

* Knee locking or trauma leading to acute surgery.
* One of the following associated injuries on the index knee:

  1. A symptomatic partial ACL rupture or any total ACL rupture determined by clinical examination (positive Lachman test and/or positive Pivot Shift) and shown on MRI;
  2. A complete Posterior Cruciate Ligament (PCL) injury;
  3. Cartilage change down to bone; grade 4 of the Kellgren Lawrence Grading Scale for Osteoarthritis visualized on X-ray;
  4. An injury to the lateral/posterolateral ligament complex with significantly increased laxity.
* A history of knee surgery other than diagnostic arthroscopy on the index knee.
* Tumors on MRI suspected for a malignancy.
* Obese patients with Body Mass Index (BMI) > 35.
* ASA 4-5 patients which can severely interfere with rehabilitation.
* General disease that effects physical function or systemic medication/abuse of steroids (e.g., rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout, pseudogout)
* Any other medical condition or treatment interfering with the completion or assessment of the trial, e.g. contraindications to MRI or surgery.
* Drugs or alcohol abuse.
* Patients unable to speak or read Dutch.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee 'Subjective Knee Form' | 3, 6, 12, 24 and 60 months
  Primary outcome will be change in physical function from baseline to 2 years measured by the International Knee Documentation Committee (IKDC) 'Subjective Knee Form', which has been validated for meniscal injuries.
  In addition, 1) the investigators will perform an economic analysis alongside the Randomized Controlled Trial (RCT) from a societal perspective and a budget impact analysis from societal, government and insurer perspective.
  2) The primary outcome after 5 years will be investigated

SECONDARY OUTCOMES:
RAND-36 Physical Functional Status Scale | 3, 6, 12 and 24 months
EQ-5D-5L Quality of life measure | 3, 6, 9, 12, 18, 24 and 60 months
Tegner Activity Scale | 3, 6, 12 and 24 months
Health Care Utilization and productivity losses | 3, 6, 9, 12, 18 and 24 months
Patient Specific Complaints questionnaire | 3, 6 ,12 and 24 months
Physical Examination | 3 and 24 months
  Performance on meniscus specific physical tests, joint line tenderness and the existence of joint effusion in the knee.
VAS pain score | 3, 6, 12, 24 and 60 months
Knee Osteoarthritis Outcome Score-Physical functioning Short from (KOOS-PS) | 60 months
  for physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf W Poolman, MD PhD, Principal Investigator — Dept. Orthopaedic Surgery Onze Lieve Vrouwe Gasthuis; Arthur de Gast, MD PhD, Principal Investigator — Dept. Orthopaedic Surgery Diakonessenhuis, Utrecht; Thijs ThM van der SChoot, MD PhD, Study Chair — Dean Board of Directors Onze Lieve Vrouwe Gasthuis; Eduard LA Mutsaerts, MD PhD, Principal Investigator — Dept. of Orthopaedic Surgery Onze Lieve Vrouwe Gasthuis; Victor A van de Graaf, MD, Study Chair — Dept. of Orthopaedic Surgery Onze Lieve Vrouwe Gasthuis; Gino MM Kerkhoffs, MD PhD, Principal Investigator — Dept. of Orthopaedic Surgery Academic Medical Center University of Amsterdam; Julius Wolkenfelt, MD, Principal Investigator — Dept. of Orthopaedic Surgery St. Lucas Andreas Hospital; Maurits W van Tulder, professor, Study Director — Professor of Health Technology Assessment Dept. Health Sciences VU University Amsterdam; Vanessa AB Scholtes, PhD, Study Director — Research coordinator Dept. of Orthopaedic Surgery Onze Lieve Vrouwe Gasthuis; Nienke Wolterbeek, PhD, Study Director — Research coordinator Dept. of Orthopaedic Surgery St. Antonius Hospital; Camille Neeter, PhD, Study Director — Neeter Physiotherapy Amsterdam; Ewoud RA van Arkel, MD PhD, Principal Investigator — Dept. of Orthopaedic Surgery MC Haaglanden
Locations (10):
- Netherlands (10):
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - St Lucas Andreas Hospital, Amsterdam, North Holland
  - Medisch Centrum Jan van Goyen, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Academic Medical Center University of Amsterdam, Amsterdam, North Holland
  - Slotervaart Ziekenhuis, Amsterdam
  - Tergooi Ziekenhuis, Hilversum
  - Medisch Centrum Haaglanden, The Hague
  - Sint Elisabeth Hospital, Tilburg
  - Diakonessenhuis, Utrecht

REFERENCES:
- [Derived] Noorduyn JCA, van de Graaf VA, Willigenburg NW, Scholten-Peeters GGM, Kret EJ, van Dijk RA, Buchbinder R, Hawker GA, Coppieters MW, Poolman RW; ESCAPE Research Group. Effect of Physical Therapy vs Arthroscopic Partial Meniscectomy in People With Degenerative Meniscal Tears: Five-Year Follow-up of the ESCAPE Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220394. doi: 10.1001/jamanetworkopen.2022.20394. PMID 35802374
- [Derived] Noorduyn JCA, Glastra van Loon T, van de Graaf VA, Willigenburg NW, Butter IK, Scholten-Peeters GGM, Coppieters MW, Poolman RW; ESCAPE Research Group; Scholtes VAB, Mutsaerts ELAR, Krijnen MR, Moojen DJF, van Deurzen DFP, Bloembergen CH, Wolkenfelt J, de Gast A, Snijders T, Saris DBF, Wolterbeek N, Neeter C, Kerkhoffs GMMJ, Peters RW, van den Brand ICJB, de Vos-Jakobs S, Spoor AB, Gosens T, Rezaie W, Hofstee DJ, Burger BJ, Haverkamp D, Vervest AMJS, van Rheenen TA, Wijsbek AE, van Arkel ERA, Thomassen BJW, Sprague S, van Tulder MW, Schavemaker M, van Dijk R, van der Kraan J. Functional Outcomes of Arthroscopic Partial Meniscectomy Versus Physical Therapy for Degenerative Meniscal Tears Using a Patient-Specific Score: A Randomized Controlled Trial. Orthop J Sports Med. 2020 Oct 29;8(10):2325967120954392. doi: 10.1177/2325967120954392. eCollection 2020 Oct. PMID 33195707
- [Derived] van de Graaf VA, van Dongen JM, Willigenburg NW, Noorduyn JCA, Butter IK, de Gast A, Saris DBF, van Tulder MW, Poolman RW; ESCAPE Research Group. How do the costs of physical therapy and arthroscopic partial meniscectomy compare? A trial-based economic evaluation of two treatments in patients with meniscal tears alongside the ESCAPE study. Br J Sports Med. 2020 May;54(9):538-545. doi: 10.1136/bjsports-2018-100065. Epub 2019 Jun 21. PMID 31227493
- [Derived] van de Graaf VA, Noorduyn JCA, Willigenburg NW, Butter IK, de Gast A, Mol BW, Saris DBF, Twisk JWR, Poolman RW; ESCAPE Research Group. Effect of Early Surgery vs Physical Therapy on Knee Function Among Patients With Nonobstructive Meniscal Tears: The ESCAPE Randomized Clinical Trial. JAMA. 2018 Oct 2;320(13):1328-1337. doi: 10.1001/jama.2018.13308. PMID 30285177
- [Derived] van de Graaf VA, Scholtes VA, Wolterbeek N, Noorduyn JC, Neeter C, van Tulder MW, Saris DB, de Gast A, Poolman RW; Escape Research Group. Cost-effectiveness of Early Surgery versus Conservative Treatment with Optional Delayed Meniscectomy for Patients over 45 years with non-obstructive meniscal tears (ESCAPE study): protocol of a randomised controlled trial. BMJ Open. 2016 Dec 21;6(12):e014381. doi: 10.1136/bmjopen-2016-014381. PMID 28003302

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT01850719/SAP_000.pdf